CLINICAL TRIAL: NCT04082273
Title: A Single Center, Randomized Control Study to Compare Efficacy and Safety of Femto-laser Created Clear Corneal Incisions with Manually Created Clear Corneal Incisions During Cataract Surgery
Brief Title: Comparison of Femto-laser and Manually Created Clear Corneal Incisions During Cataract Surgery
Acronym: Z8_CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPFEM-0005-CH
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2021-07

CONDITIONS: Cataract
Keywords: Induced corneal Astigmatism; Clear corneal incisions; Femto-laser
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Femtosecond Laser for Cataract Surgery (Experimental): Capsulotomy, lens fragmentation and Clear Corneal Incisions with FEMTO LDV Z8, followed by ultrasound phacoemulsification and IOL implantation.
  Interventions: Device: Femtosecond Laser for Cataract Surgery
- Conventional Cataract Surgery (Active Comparator): Clear Corneal Incisions, conventional capsulorhexis and ultrasound phacoemulsification and IOL implantation. Control treatment where the clear corneal incisions and capsulorhexis are performed manually and the lens fragmentation is performed with the phacoemulsification device.
  Interventions: Other: Conventional Cataract Surgery

INTERVENTIONS:
Device: Femtosecond Laser for Cataract Surgery — Cataract Surgery on study eye according to conventional procedure, with the exception of three steps (Capsulotomy, Lens Fragmentation and Clear Corneal Incisions) which are performed with a Femtosecond Laser in the laser treatment group. Equipment uesd for measurements is the same for both groups and in line with the normal equipment used for the conventional cataract treatment
  Arms: Femtosecond Laser for Cataract Surgery
Other: Conventional Cataract Surgery — Cataract surgery will be performed conventionally, this means the clear corneal incisions will be performed manually by a blade, the capsulorhexis will be performed manually by a hook, and the lens extraction will be done by phacoemulsification
  Arms: Conventional Cataract Surgery

SUMMARY:
The aim of this study is to test the hypothesis, that in terms of Surgically Induced corneal Astigmatism (SIA), Higher-order Aberrations (HOA), and wound geometry the femtosecond clear corneal incisions (CCIs) created during cataract surgery are not inferior when compared to manual CCIs.

The potential risks associated with application of the femtosecond laser in this study are no greater or in most cases less than those associated with the standard manual cataract surgical procedure, and the potential benefits (such as precision and reproducibility) are greater than with the standard manual cataract surgery. Therefore, the risk-to-benefit ratio is very low, such that the potential benefits for a subject participating in this study exceed the potential risks

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens implantation
* Able to co-operate with the docking system for the femtosecond laser
* Clear corneal media
* 40 years of age or older
* Willing and able to return for scheduled follow-up examinations

Exclusion Criteria:

* Minimal and maximal K-values of the central 3mm zone that differ by more than 5D on a keratometric map of the cornea
* Maximum K-value that exceeds 58.D
* Minimal K-value of less than 37.D
* Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
* Poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Manifest Glaucoma+OHT (ocular hypertension), pseudoexfoliation
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye
* Known sensitivity to planned concomitant medications
* History of lens or zonular instability
* Keratoconus or keratectasia
* Immune compromised or diagnosis of connective tissue disease, clinically significant atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, RA, collagenosis and other acute or chronic illnesses that increases the risk to the subject or confounds the outcomes of this study, in the opinion of the study Pl.
* Anterior chamber depth (ACD) < 1.5 mm or ACD > 4.8 mm as measured from the corneal endothelium.
* Extensive corneal scarring, pterygium
* Developmental disability or cognitive impairment (would preclude adequate comprehension of the IC form and/or the ability to record the study measurements)
* Concurrent participation in another ophthalmological clinical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline (pre-operative) Surgically Induced corneal Astigmatism (SIA) measured by means of corneal topography Galilei G2 | Baseline = Pre-operative, Follow-up = 12 days, 4 weeks and 6 weeks after surgery

SECONDARY OUTCOMES:
Change from baseline (pre-operative) Higher-order aberrations (HOAs) by means of aberrometry using Galilei G2 | Baseline = Pre-operative, Follow-up = 12 days, 4 weeks and 6 weeks after surgery
Central corneal thickness (CCT) | Baseline = Pre-operative, Follow-up = 1 day, 12 days, 4 weeks and 6 weeks after surgery
Endothelial cell density (ECD) | Baseline = Pre-operative, Follow-up = 1 day, 12 days, 4 weeks and 6 weeks after surgery
Effective Phacoemulsification Time (EPT) | Baseline = Treatment day
Ultrasound total time (US) | Baseline = Treatment day
Achieved CCI architecture | 1 day postoperative and 12 days postoperative
  Presence of Descemet membrane detachment, posterior and anterior wound gape, if present size) will be analyzed on OCT images
Intra- and post-operative CCI related complications rate | Baseline = Treatment day, Follow-up = 1 day, 12 days, 4 weeks and 6 weeks after surgery
FEMTO LDV Z8 OCT auto - detection accuracy | Baseline = Treatment day
  Analyzed on intra-operative Z8 OCT images

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Pajic, MD, PhD, Principal Investigator — Augenklinik ORASIS AG
Locations (1):
- Augenklinik ORASIS AG, Reinach, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brian G, Taylor H. Cataract blindness--challenges for the 21st century. Bull World Health Organ. 2001;79(3):249-56. Epub 2003 Jul 7. PMID 11285671
- [Background] Nagy Z, Takacs A, Filkorn T, Sarayba M. Initial clinical evaluation of an intraocular femtosecond laser in cataract surgery. J Refract Surg. 2009 Dec;25(12):1053-60. doi: 10.3928/1081597X-20091117-04. PMID 20000286
- [Background] He L, Sheehy K, Culbertson W. Femtosecond laser-assisted cataract surgery. Curr Opin Ophthalmol. 2011 Jan;22(1):43-52. doi: 10.1097/ICU.0b013e3283414f76. PMID 21150606
- [Background] Trikha S, Turnbull AM, Morris RJ, Anderson DF, Hossain P. The journey to femtosecond laser-assisted cataract surgery: new beginnings or a false dawn? Eye (Lond). 2013 Apr;27(4):461-73. doi: 10.1038/eye.2012.293. Epub 2013 Feb 1. PMID 23370418
- [Background] Chang JS, Chen IN, Chan WM, Ng JC, Chan VK, Law AK. Initial evaluation of a femtosecond laser system in cataract surgery. J Cataract Refract Surg. 2014 Jan;40(1):29-36. doi: 10.1016/j.jcrs.2013.08.045. Epub 2013 Nov 22. PMID 24269139
- [Background] Grewal DS, Basti S. Comparison of morphologic features of clear corneal incisions created with a femtosecond laser or a keratome. J Cataract Refract Surg. 2014 Apr;40(4):521-30. doi: 10.1016/j.jcrs.2013.11.028. Epub 2014 Feb 22. PMID 24568722
- [Background] Baig NB, Cheng GP, Lam JK, Jhanji V, Chong KK, Woo VC, Tham CC. Intraocular pressure profiles during femtosecond laser-assisted cataract surgery. J Cataract Refract Surg. 2014 Nov;40(11):1784-9. doi: 10.1016/j.jcrs.2014.04.026. Epub 2014 Sep 24. PMID 25261391
- [Background] Reddy KP, Kandulla J, Auffarth GU. Effectiveness and safety of femtosecond laser-assisted lens fragmentation and anterior capsulotomy versus the manual technique in cataract surgery. J Cataract Refract Surg. 2013 Sep;39(9):1297-306. doi: 10.1016/j.jcrs.2013.05.035. PMID 23988242
- [Background] Nagy ZZ, Kranitz K, Takacs AI, Mihaltz K, Kovacs I, Knorz MC. Comparison of intraocular lens decentration parameters after femtosecond and manual capsulotomies. J Refract Surg. 2011 Aug;27(8):564-9. doi: 10.3928/1081597X-20110607-01. Epub 2011 Jun 20. PMID 21688765
- [Background] Friedman NJ, Palanker DV, Schuele G, Andersen D, Marcellino G, Seibel BS, Batlle J, Feliz R, Talamo JH, Blumenkranz MS, Culbertson WW. Femtosecond laser capsulotomy. J Cataract Refract Surg. 2011 Jul;37(7):1189-98. doi: 10.1016/j.jcrs.2011.04.022. PMID 21700099
- [Background] Palanker DV, Blumenkranz MS, Andersen D, Wiltberger M, Marcellino G, Gooding P, Angeley D, Schuele G, Woodley B, Simoneau M, Friedman NJ, Seibel B, Batlle J, Feliz R, Talamo J, Culbertson W. Femtosecond laser-assisted cataract surgery with integrated optical coherence tomography. Sci Transl Med. 2010 Nov 17;2(58):58ra85. doi: 10.1126/scitranslmed.3001305. PMID 21084720
- [Background] Pajic B, Vastardis I, Gatzioufas Z, Pajic-Eggspuehler B. First experience with the new high-frequency femtosecond laser system (LDV Z8) for cataract surgery. Clin Ophthalmol. 2014 Dec 8;8:2485-9. doi: 10.2147/OPTH.S72983. eCollection 2014. PMID 25525326
- [Background] Abell RG, Kerr NM, Vote BJ. Femtosecond laser-assisted cataract surgery compared with conventional cataract surgery. Clin Exp Ophthalmol. 2013 Jul;41(5):455-62. doi: 10.1111/ceo.12025. Epub 2012 Dec 10. PMID 23078347
- [Background] Ferreira TB, Ribeiro FJ, Pinheiro J, Ribeiro P, O'Neill JG. Comparison of Surgically Induced Astigmatism and Morphologic Features Resulting From Femtosecond Laser and Manual Clear Corneal Incisions for Cataract Surgery. J Refract Surg. 2018 May 1;34(5):322-329. doi: 10.3928/1081597X-20180301-01. PMID 29738588
- [Background] Liu YC, Wilkins M, Kim T, Malyugin B, Mehta JS. Cataracts. Lancet. 2017 Aug 5;390(10094):600-612. doi: 10.1016/S0140-6736(17)30544-5. Epub 2017 Feb 25. PMID 28242111
- [Background] Olson RJ, Braga-Mele R, Chen SH, Miller KM, Pineda R 2nd, Tweeten JP, Musch DC. Cataract in the Adult Eye Preferred Practice Pattern(R). Ophthalmology. 2017 Feb;124(2):P1-P119. doi: 10.1016/j.ophtha.2016.09.027. Epub 2016 Oct 13. No abstract available. PMID 27745902